CLINICAL TRIAL: NCT05307705
Title: A Study of LOXO-783 Administered as Monotherapy and in Combination With Anticancer Therapies for Patients With Advanced Breast Cancer and Other Solid Tumors With a PIK3CA H1047R Mutation
Brief Title: A Study of LOXO-783 in Patients With Breast Cancer/Other Solid Tumors
Acronym: PIKASSO-01
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18394; 2022-000175-40 (EudraCT Number); J4C-OX-JZUA (Other: Eli Lilly and Company); LOXO-PIK-21001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-03-25; First posted 2022-04-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Imlunestrant; abemaciclib; Anastrozole; exemestane; Letrozole; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1A: LOXO-783 Monotherapy Dose Escalation (Experimental): LOXO-783 administered orally
  Interventions: Drug: LOXO-783
- Phase 1B: Part A (Experimental): LOXO-783 administered orally in combination with fulvestrant intramuscularly, imlunestrant orally, or an aromatase inhibitor orally
  Interventions: Drug: LOXO-783; Drug: Fulvestrant; Drug: Imlunestrant; Drug: Anastrozole, Exemestane, or Letrozole
- Phase 1B: Part B (Experimental): LOXO-783 orally in combination with abemaciclib and either physician's choice aromatase inhibitor orally, fulvestrant intramuscularly, or imlunestrant orally
  Interventions: Drug: LOXO-783; Drug: Fulvestrant; Drug: Imlunestrant; Drug: Abemaciclib; Drug: Anastrozole, Exemestane, or Letrozole
- Phase 1B: Part C (Experimental): LOXO-783 orally in combination with fulvestrant intramuscularly
  Interventions: Drug: LOXO-783; Drug: Fulvestrant
- Phase 1B: Part D (Experimental): LOXO-783 orally in combination with paclitaxel intravenously
  Interventions: Drug: LOXO-783; Drug: Paclitaxel
- Phase 1B: Part E (Experimental): LOXO-783 orally
  Interventions: Drug: LOXO-783
- Phase 1B: Part F (Experimental): Multiple randomized dose levels of LOXO-783 orally with fulvestrant intramuscularly
  Interventions: Drug: LOXO-783; Drug: Fulvestrant

INTERVENTIONS:
Drug: LOXO-783 — Oral
  Other Names: LY3849524
Drug: Fulvestrant — Intramuscular
  Arms: Phase 1B: Part A; Phase 1B: Part B; Phase 1B: Part C; Phase 1B: Part F
Drug: Imlunestrant — Oral
  Other Names: LY3484356
  Arms: Phase 1B: Part A; Phase 1B: Part B
Drug: Abemaciclib — Oral
  Other Names: LY2835219
  Arms: Phase 1B: Part B
Drug: Anastrozole, Exemestane, or Letrozole — Oral
  Arms: Phase 1B: Part A; Phase 1B: Part B
Drug: Paclitaxel — Intravenous
  Arms: Phase 1B: Part D

SUMMARY:
The main purpose of this study is to learn more about the safety, side effects, and effectiveness of LOXO-783. LOXO-783 may be used to treat breast cancer and other solid tumors that have a change in a particular gene (known as the PIK3CA gene). Participation could last up to 36 months (3 years) and possibly longer if the disease does not get worse.

ELIGIBILITY:
Inclusion Criteria:

* Have advanced breast cancer or another solid tumor with the presence of a phosphatidylinositol 3-kinase catalytic subunit alpha (PIK3CA) H1047R mutation (or other Sponsor and safety review committee (SRC)-approved, activating PIK3CA mutations other than H1047R mutation)
* Have adequate archival tumor tissue sample available or be approved by the Sponsor for enrollment if no tumor sample is available.
* Have stopped all cancer treatment and have recovered from the major side effects
* Have adequate organ function, as measured by blood tests
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Patients must have

  * Measurable disease

    --- Patients with non-breast tumor types must have at least 1 measurable lesion
  * Non-measurable bone disease (at least 1 bone lesion in breast cancer patients only)
* For patients with an estrogen receptor (ER)+ breast cancer diagnosis:

  * If female, must be postmenopausal
  * If male, must agree to use hormone suppression
* Phase 1a:

  -- Dose escalation and backfill patients:
  * Advanced solid tumor
  * Patients may have had up to 5 prior regimens for advanced disease
* Phase 1b:

  * Part A:

    * ER+/human epidermal growth factor receptor 2 (HER2)- advanced breast cancer
    * Patients may have had up to 5 prior regimens for advanced disease ---- Prior cyclin dependent kinase (CDK)4/6 inhibitor therapy required
  * Part B:

    * ER+/HER2- advanced breast cancer
    * Patients may have had up to 2 prior regimens for advanced disease.
  * Part C:

    * ER+/HER2- advanced breast cancer
    * Patients may have had up to 5 prior regimens for advanced disease.

      ---- Prior CDK4/6 inhibitor therapy required.
    * Have a diagnosis of diabetes mellitus Type 2
  * Part D:

    * Advanced breast cancer
    * Patients may have had up to 5 prior regimens for advanced disease.
  * Part E:

    * Advanced solid tumor
    * Patients may have had up to 3 prior regimens for advanced disease advanced disease
  * Part F:

    * ER+/HER2- advanced breast cancer
    * Patients may have had up to 5 prior regimens for advanced disease

      * Prior cyclin dependent kinase (CDK)4/6 inhibitor therapy required

Exclusion Criteria:

* Medical Conditions

  * Colorectal cancer
  * Endometrial cancers with specific concurrent oncogenic alterations
  * A history of known active or suspected

    * Diabetes mellitus Type 1 or
    * Diabetes mellitus Type 2 requiring antidiabetic medication (Phase 1a and all parts of Phase 1b except Part C).
    * Serious concomitant systemic disorder
* Known or suspected history of untreated or uncontrolled central nervous system (CNS) involvement.
* Active uncontrolled systemic bacterial, viral, fungal, or parasitic infection, or other clinically significant active disease process
* Prior exposure to phosphatidylinositol 3-kinase/protein kinase B/mammalian target of rapamycin (PI3K/AKT/mTOR) inhibitor(s), except in certain circumstances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1 a: To determine the maximum tolerated dose/recommended phase 2 dose (MTD/RP2D) of LOXO-783: Number of patients with dose-limiting toxicities (DLTs) | During the first 28-day cycle of LOXO-783 treatment
  Number of patients with DLTs
Phase 1 a: To determine the MTD/RP2D of LOXO-783: Number of patients with DLT-equivalent toxicities | During the first 28-day cycle of LOXO-783 treatment
  Number of patients with DLT-equivalent toxicities

SECONDARY OUTCOMES:
To assess the pharmacokinetics (PK) of LOXO-783: Area under the concentration versus time curve (AUC) | Up to 2 months
  PK of LOXO-783: AUC
To assess the PK of LOXO-783: Maximum drug concentration (Cmax) | Up to 2 months
  PK of LOXO-783: Cmax
To evaluate the preliminary antitumor activity of LOXO-783: Overall response rate (ORR) | Up to approximately 36 months or 3 years
  ORR per investigator assessed Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)
To evaluate the preliminary antitumor activity of LOXO-783: Best overall response (BOR) | Up to approximately 36 months or 3 years
  BOR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LOXO-783: Duration of response (DOR) | Up to approximately 36 months or 3 years
  DOR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LOXO-783: Disease control rate (DCR) | Up to approximately 36 months or 3 years
  DCR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LOXO-783: Clinical benefit rate (CBR) | Up to approximately 36 months or 3 years
  CBR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LOXO-783: Time to response (TTR) | Up to approximately 36 months or 3 years
  TTR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LOXO-783: Progression free survival (PFS) | Up to approximately 36 months or 3 years
  PFS per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LOXO-783: Overall survival (OS) | Up to approximately 36 months or 3 years
  OS per investigator assessed RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (50):
- United States (17):
  - Mayo Clinic of Scottsdale, Scottsdale, Arizona
  - UCLA Medical Center, Los Angeles, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Stanford University Hospital, Stanford, California
  - Mayo Clinic, Jacksonville, Florida
  - Winship Cancer Center Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wilmot Cancer Institute, Rochester, New York
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
- Australia (3):
  - Cancer Research SA, Adelaide
  - Peter Maccallum Cancer Institute Erb, East Melbourne
  - St Vincent's Hospital, Sydney
- Belgium (2):
  - Institut Jules Bordet, Anderlecht
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Canada (2):
  - Princess Margaret Hospital (Hong Kong), Toronto
  - BC Cancer Vancouver, Vancouver
- China (3):
  - Beijing Cancer hospital, Beijing
  - The Third Hospital of Nanchang, Nanchang
  - Fudan University Shanghai Cancer Center, Shanghai
- France (5):
  - Centre Leon Berard, Lyon
  - Institut Curie, Paris
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - ICANS_Institut de Cancerologie Strasbourg Europe, Strasbourg
  - Gustave Roussy, Villejuif
- Universitätsklinikum Erlangen, Erlangen, Germany
- Japan (4):
  - National Cancer Center Hospital, Chūōku
  - The Cancer Institute Hospital of JFCR, Kōtō City
  - Kyoto University Hospital, Kyoto
  - Aichi Cancer Center Hospital, Nagoya
- National Cancer Centre Singapore, Singapore, Singapore
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (8):
  - Hospital Universitario Quiron Dexeus, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova Valencia, Valencia
- United Kingdom (2):
  - Royal Marsden NHS Trust, London
  - Royal Marsden Hospital (Sutton), Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LOXO-783 in Patients With Breast Cancer/Other Solid Tumors — https://trials.lilly.com/en-US/trial/338185